CLINICAL TRIAL: NCT03158844
Title: HIV Care Cascade and Linkage to Antiretroviral Therapy Among Hospitalized Adults in Lusaka, Zambia
Acronym: COLAH
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University Teaching Hospital (Unknown); Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Principal Investigator, Michael Vinikoor, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: F160812007
Record Dates: First submitted 2017-05-08; First posted 2017-05-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2018-08

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood will be drawn via phlebotomy for patients for whom CD4 and HIV viral load results are not available at baseline. For participants that have initiated ART treatment, we will collect a dried blood spot card using 5 drops of blood from finger prick to measure viral load 90 days after discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HIV+ patients (Standard of care): 300 HIV-infected and hospitalized adult patients at the University Teaching Hospital (UTH) will be recruited.
  Interventions: Other: Standard of care
- Health systems informants: 15 key Zambian health systems informants and leaders who can discuss inpatient care and the process of linking hospitalized patients to HIV care.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Routine standard of care per Ministry of Health protocol, including blood draws and examinations.

SUMMARY:
The population of inpatients is large in Zambia; however, because of poor linkages between hospitals and community HIV care, there are few data to analyze their engagement in HIV care before and after hospitalization. The goal of the study is to learn more about Zambian adults who are HIV-infected and get hospitalized. The purpose of this study is to gather formative, preliminary data, to be used in future grant applications to improve linkage and engagement in HIV care in Zambia.

DETAILED DESCRIPTION:
The main objective of this study is to generate preliminary data on the outcomes of Zambian HIV-infected individuals after discharge from University Teaching Hospital (UTH) Internal Medicine wards which can inform development of a linkage intervention. Our central hypothesis is that in Sub-Saharan African settings like Zambia hospitalizations among HIV-infected individuals are driven by suboptimal linkage and initiation of ART following HIV diagnosis. Specific Aims: (a) Characterize the distribution of hospitalized 300 HIV-infected adults across the HIV care continuum. (b) Identify structural, psychosocial, clinic, and medical factors that predict suboptimal linkage to care and ART initiation after 90 days of hospital discharge among HIV-infected Zambians.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* HIV-infected as documented in the UTH file
* Admitted to Internal Medicine Ward at UTH

Exclusion Criteria:

* Unable to provide informed consent
* Not planning to remain in Lusaka province for 3 months after discharge

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In part 1, people will be recruited in a random fashion from HIV-infected patients hospitalized at the University Teaching Hospital (UTH) as documented in their UTH medical file regardless of their HIV treatment status. The bed spaces in the wards will be enumerated and using a random number generator the team will select patients for screening for study inclusion.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Undetectable HIV viral load at 90 days post-discharge | 90 days after hospital discharge
  Numerator is number with HIV RNA <1000 c/mL tested at 90 days after hospital discharge; denominator is the # enrolled

SECONDARY OUTCOMES:
Proportion of HIV-infected inpatients who are on ART upon admission | Baseline
  Numerator is number who report taking ART up to the time of admission; denominator is the # enrolled
Mortality rate | 90 days after hospital discharge
  Mortality from time of enrollment to 90 days after discharge
ART initiation | Baseline and 90 days after hospital discharge
  Proportion not on ART upon admission to hospital who are on ART at 90 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Vinikoor, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided